CLINICAL TRIAL: NCT00687804
Title: A Randomized, Double-masked, Multicenter, Laser-controlled Phase III Study Assessing the Efficacy and Safety of Ranibizumab (Intravitreal Injections) as Adjunctive and Mono-therapy in Patients With Visual Impairment Due to Diabetic Macular Edema
Brief Title: A 12 Month Core Study to Assess the Efficacy and Safety of Ranibizumab (Intravitreal Injections) in Patients With Visual Impairment Due to Diabetic Macular Edema and a 24 Month Open-label Extension Study
Acronym: RESTORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRFB002D2301; EUDRACT: 2007-004877-24; NCT00906464 (obsolete NCT alias)
Record Dates: First submitted 2008-05-27; First posted 2008-06-02 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Diabetic Macular Edema
Keywords: DME; Diabetic; macula; edema; ranibizumab; RESTORE
MeSH Terms: conditions — Edema | interventions — Ranibizumab; Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Ranibizumab 0.5 mg (Experimental): Ranibizumab 0.5 mg was administered monthly by intravitreal injection in the study eye for 3 months. After the third injection, treatment was suspended if either one of the following criteria was met:
  Improvement in best corrected visual acuity (BCVA) could not be attributed to treatment at the last 2 visits, in the opinion of the investigator, or BCVA > 84 letters (approximate Snellen equivalent of 20/20) was observed at the last 2 last visits.
  Patients also received sham laser treatment on Day 1 and subsequently at intervals of at least 3 months, if deemed necessary by the evaluating physician.
  Active/sham laser treatment was always administered before (sham) intravitreal injections. The minimum interval between the 2 treatments was 30 minutes.
  In the extension study at the investigator's discretion, patients received open-label ranibizumab 0.5 mg intravitreal injections once a month until stable vision was reached (a maximum of 24 injections) and could receive laser therapy.
  Interventions: Drug: Ranibizumab; Procedure: Laser; Procedure: Sham laser
- Ranibizumab 0.5 mg + laser (Experimental): Ranibizumab 0.5 mg was administered monthly by intravitreal injection in the study eye for 3 months. After the third injection, treatment was suspended if either one of the following criteria was met:
  Improvement in best corrected visual acuity (BCVA) could not be attributed to treatment at the last 2 visits, in the opinion of the investigator, or BCVA > 84 letters (approximate Snellen equivalent of 20/20) was observed at the last 2 last visits.
  Patients also received active laser treatment on Day 1 and subsequently at intervals of at least 3 months, if deemed necessary by the evaluating physician.
  Active/sham laser treatment was always administered before (sham) intravitreal injections. The minimum interval between the 2 treatments was 30 minutes.
  In the extension study at the investigator's discretion, patients received open-label ranibizumab 0.5 mg intravitreal injections once a month until stable vision was reached (a maximum of 24 injections) and could receive laser therapy.
  Interventions: Drug: Ranibizumab; Procedure: Laser
- Laser (Active Comparator): Laser photocoagulation treatment was administered on Day 1 and at intervals of at least 3 months, if deemed necessary by the physician. Patients also received monthly sham intravitreal injection in the study eye for 3 consecutive months. After the third injection, treatment was suspended if either one of the following criteria was met:
  Improvement in best corrected visual acuity (BCVA) could not be attributed to treatment at the last 2 visits, in the opinion of the investigator, or BCVA > 84 letters (approximate Snellen equivalent of 20/20) was observed at the last 2 last visits.
  Active/sham laser treatment was always administered before (sham) intravitreal injections. The minimum interval between the 2 treatments was 30 minutes.
  In the extension study at the investigator's discretion, patients received open-label ranibizumab 0.5 mg intravitreal injections once a month until stable vision was reached (a maximum of 24 injections) and could receive laser therapy.
  Interventions: Drug: Ranibizumab; Procedure: Laser; Drug: Sham to ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.5 mg ranibizumab administered by intravitreal injection.
Procedure: Laser — Laser photocoagulation treatment
Procedure: Sham laser — Sham to laser procedure.
  Arms: Ranibizumab 0.5 mg
Drug: Sham to ranibizumab — Sham to ranibizumab administered as an intravitreal injection.
  Arms: Laser

SUMMARY:
CRFB002D2301: The core study was designed to confirm the efficacy and safety of ranibizumab (0.5 mg) as adjunctive therapy when added to laser photocoagulation and/or mono-therapy in patients with visual impairment due to diabetic macular edema.

CRFB002D2301E1: A 24 month open-label extension study for participants who completed the 12 month core study evaluated the long-term safety and efficacy of ranibizumab (0.5 mg) as symptomatic treatment for visual impairment due to diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity impairment
* Diabetic macular edema in at least one eye
* Type 1 or type 2 diabetes mellitus
* Medication for the diabetes treatment must be stable for the last 3 months

Exclusion Criteria:

* Patients with uncontrolled systemic or ocular diseases
* Laser photocoagulation in the study eye for the last 3 months
* Any history of any intraocular surgery in the study eye within the past 3 months
* Blood pressure > 160/100 mmHg

Extension Inclusion Criteria:

-Completion of the Core Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Novartis Investigative Site, Melbourne, Australia
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Ontario, Canada
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Düsseldorf, Germany
- Novartis Investigative Site, Athens, Greece
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Florence, Italy
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Barcelona, Spain
- Novartis Investigational Site, Zurich, Switzerland
- Novartis Investigative Site, Ankara, Turkey (Türkiye)
- Novartis Investigative Site, Upton, United Kingdom

REFERENCES:
- [Derived] Bressler NM, Varma R, Mitchell P, Suner IJ, Dolan C, Ward J, Ferreira A, Ehrlich JS, Turpcu A. Effect of Ranibizumab on the Decision to Drive and Vision Function Relevant to Driving in Patients With Diabetic Macular Edema: Report From RESTORE, RIDE, and RISE Trials. JAMA Ophthalmol. 2016 Feb;134(2):160-6. doi: 10.1001/jamaophthalmol.2015.4636. PMID 26584450
- [Derived] Mitchell P, Massin P, Bressler S, Coon CD, Petrillo J, Ferreira A, Bressler NM. Three-year patient-reported visual function outcomes in diabetic macular edema managed with ranibizumab: the RESTORE extension study. Curr Med Res Opin. 2015 Nov;31(11):1967-75. doi: 10.1185/03007995.2015.1081880. Epub 2015 Oct 6. PMID 26327116
- [Derived] Bressler NM, Varma R, Suner IJ, Dolan CM, Ward J, Ehrlich JS, Colman S, Turpcu A; RIDE and RISE Research Groups. Vision-related function after ranibizumab treatment for diabetic macular edema: results from RIDE and RISE. Ophthalmology. 2014 Dec;121(12):2461-72. doi: 10.1016/j.ophtha.2014.07.008. Epub 2014 Aug 20. PMID 25148789
- [Derived] Schmidt-Erfurth U, Lang GE, Holz FG, Schlingemann RO, Lanzetta P, Massin P, Gerstner O, Bouazza AS, Shen H, Osborne A, Mitchell P; RESTORE Extension Study Group. Three-year outcomes of individualized ranibizumab treatment in patients with diabetic macular edema: the RESTORE extension study. Ophthalmology. 2014 May;121(5):1045-53. doi: 10.1016/j.ophtha.2013.11.041. Epub 2014 Feb 1. PMID 24491642
- [Derived] Mitchell P, Bressler N, Tolley K, Gallagher M, Petrillo J, Ferreira A, Wood R, Bandello F; RESTORE Study Group. Patient-reported visual function outcomes improve after ranibizumab treatment in patients with vision impairment due to diabetic macular edema: randomized clinical trial. JAMA Ophthalmol. 2013 Oct;131(10):1339-47. doi: 10.1001/jamaophthalmol.2013.4592. PMID 23974915
- [Derived] Mitchell P, Bandello F, Schmidt-Erfurth U, Lang GE, Massin P, Schlingemann RO, Sutter F, Simader C, Burian G, Gerstner O, Weichselberger A; RESTORE study group. The RESTORE study: ranibizumab monotherapy or combined with laser versus laser monotherapy for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):615-25. doi: 10.1016/j.ophtha.2011.01.031. PMID 21459215

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the 12 month randomized core study CRFB002D2301 were eligible to participate in the 24 month open-label extension study CRFB002D2301E1. The reporting groups for the participants in the extension study are according to their assigned treatment groups in the core study.
Groups:
- Ranibizumab 0.5 mg + Laser: Ranibizumab 0.5 mg was administered monthly by intravitreal injection in the study eye for 3 months. After the third injection, treatment was suspended if either one of the following criteria was met:
  Improvement in best corrected visual acuity (BCVA) could not be attributed to treatment at the last 2 visits, in the opinion of the investigator, or BCVA > 84 letters (approximate Snellen equivalent of 20/20) was observed at the last 2 last visits.
  Patients also received active laser treatment on Day 1 and subsequently at intervals of at least 3 months, if deemed necessary by the physician.
  Active/sham laser treatment was always administered before (sham) intravitreal injections. The minimum interval between the 2 treatments was 30 minutes.
  In the extension study at the investigator's discretion, patients received open-label ranibizumab 0.5 mg intravitreal injections once a month until stable vision was reached (a maximum of 24 injections) and could receive laser therapy.
- Laser: Active laser photocoagulation treatment was administered on Day 1 and at intervals of at least 3 months, if deemed necessary by the evaluating physician. Patients also received monthly sham intravitreal injection in the study eye for 3 consecutive months. After the third injection, treatment was suspended if either one of the following criteria was met:
  Improvement in best corrected visual acuity (BCVA) could not be attributed to treatment at the last 2 visits, in the opinion of the investigator, or BCVA > 84 letters (approximate Snellen equivalent of 20/20) was observed at the last 2 last visits.
  Active/sham laser treatment was always administered before (sham) intravitreal injections. The minimum interval between the 2 treatments was 30 minutes.
  In the extension study at the investigator's discretion, patients received open-label ranibizumab 0.5 mg intravitreal injections once a month until stable vision was reached (a maximum of 24 injections) and could receive laser therapy.
Period: Core Study
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser
Started | 116 | 118 | 111
Completed | 102 | 103 | 98
Not Completed | 14 | 15 | 13
Not completed — Adverse Event | 5 | 3 | 3
Not completed — Abnormal laboratory value(s) | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 7 | 7
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Death | 2 | 2 | 2
Not completed — Protocol Violation | 1 | 1 | 0
Period: Open-Label Extension Study
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser
Started | 83 | 83 | 74
Did Not Receive Ranibizumab in Extension | 16 | 21 | 15
Completed | 73 | 72 | 63
Not Completed | 10 | 11 | 11
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Subject withdrew consent | 3 | 4 | 4
Not completed — Lost to Follow-up | 2 | 1 | 2
Not completed — Administrative problems | 1 | 1 | 0
Not completed — Death | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Ranibizumab 0.5 mg: Ranibizumab 0.5 mg was administered monthly by intravitreal injection in the study eye for 3 months. After the third injection, treatment was suspended if either one of the following criteria was met:
  Improvement in best corrected visual acuity (BCVA) could not be attributed to treatment at the last 2 visits, in the opinion of the investigator, or BCVA > 84 letters (approximate Snellen equivalent of 20/20) was observed at the last 2 last visits.
  Patients also received sham laser treatment on Day 1 and subsequently at intervals of at least 3 months, if deemed necessary by the evaluating physician.
  Active/sham laser treatment was always administered before (sham) intravitreal injections. The minimum interval between the 2 treatments was 30 minutes.
- Ranibizumab 0.5 mg + Laser: Ranibizumab 0.5 mg was administered monthly by intravitreal injection in the study eye for 3 months. After the third injection, treatment was suspended if either one of the following criteria was met:
  Improvement in best corrected visual acuity (BCVA) could not be attributed to treatment at the last 2 visits, in the opinion of the investigator, or BCVA > 84 letters (approximate Snellen equivalent of 20/20) was observed at the last 2 last visits.
  Patients also received active laser treatment on Day 1 and subsequently at intervals of at least 3 months, if deemed necessary by the evaluating physician.
  Active/sham laser treatment was always administered before (sham) intravitreal injections. The minimum interval between the 2 treatments was 30 minutes.
- Laser: Laser photocoagulation treatment was administered on Day 1 and subsequently at intervals of at least 3 months, if deemed necessary by the evaluating physician. Patients also received monthly sham intravitreal injection in the study eye for 3 consecutive months. After the third injection, treatment was suspended if either one of the following criteria was met:
  Improvement in best corrected visual acuity (BCVA) could not be attributed to treatment at the last 2 visits, in the opinion of the investigator, or BCVA > 84 letters (approximate Snellen equivalent of 20/20) was observed at the last 2 last visits.
  Active/sham laser treatment was always administered before (sham) intravitreal injections. The minimum interval between the 2 treatments was 30 minutes.
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser | Total
Number analyzed (Participants) | 116 | 118 | 111 | 345
Age Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.29) | 64.0 (8.15) | 63.5 (8.81) | 63.5 (8.75)
Age, Customized [Number; unit: Participants]
  < 55 years | 24 | 14 | 13 | 51
  55 - <65 years | 41 | 42 | 53 | 136
  65 - <75 years | 40 | 53 | 31 | 124
  >=75 years | 11 | 9 | 14 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 48 | 53 | 144
  Male | 73 | 70 | 58 | 201

OUTCOME MEASURES:

1. Primary Outcome: Core Study: Difference Between the Baseline Level of Visual Acuity (Letters) of the Study Eye and the Mean Visual Acuity Averaged Over All Monthly Post-baseline Assessments From Month 1 to Month 12
Description: Visual acuity (VA) was assessed on both eyes during every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters.
Time Frame: Baseline through the end of study (Month 12)
Population: Full analysis set consists of all patients who received at least one application of study treatment and had at least one post-baseline assessment for BCVA. Following the intent to treat principle, patients were analyzed according to the treatment assigned. Last Observation Carried Forward (LOCF) imputation was utilized.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser
Number analyzed (Participants) | 115 | 118 | 110
Letters
  Baseline | 64.7 (10.07) | 63.4 (9.99) | 62.6 (11.01)
  Average Month 1 to month 12 | 70.8 (10.53) | 69.2 (11.44) | 63.4 (12.26)
  Change from Baseline | 6.1 (6.43) | 5.9 (7.92) | 0.8 (8.56)

2. Secondary Outcome: Core Study: Categorized Change in Visual Acuity (Letters) of the Study Eye From Baseline at Month 12
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser
Number analyzed (Participants) | 115 | 118 | 110
Participants
  Gain of ≥ 10 letters | 43 | 51 | 17
  Loss of ≥ 10 letters | 4 | 5 | 14
  Gain of ≥ 15 letters | 26 | 27 | 9
  Loss of ≥ 15 letters | 1 | 4 | 9

3. Secondary Outcome: Core Study: Mean Change From Baseline in Visual Acuity (Letters) of the Study Eye Over Time
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Full analysis set, utilizing last observation carried forward.
Measure: Mean (Standard Error); unit: Letters
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser
Number analyzed (Participants) | 115 | 118 | 110
Letters
  Month 1 | 2.9 (0.49) | 3.1 (0.56) | 0.5 (0.64)
  Month 2 | 4.4 (0.64) | 4.9 (0.56) | 0.4 (0.84)
  Month 3 | 5.9 (0.65) | 5.8 (0.65) | -0.5 (0.92)
  Month 4 | 5.3 (0.68) | 5.4 (0.69) | 0.5 (0.92)
  Month 5 | 5.9 (0.68) | 5.7 (0.76) | 0.9 (0.88)
  Month 6 | 6.7 (0.68) | 6.2 (0.78) | 0.9 (0.94)
  Month 7 | 7.0 (0.72) | 6.5 (0.84) | 1.1 (0.98)
  Month 8 | 7.1 (0.75) | 6.4 (1.06) | 1.3 (0.96)
  Month 9 | 6.8 (0.76) | 6.8 (1.05) | 1.4 (0.90)
  Month 10 | 7.3 (0.77) | 6.4 (1.04) | 0.8 (1.00)
  Month 11 | 6.9 (0.79) | 6.8 (1.10) | 1.4 (0.95)
  Month 12 | 6.8 (0.77) | 6.4 (1.08) | 0.9 (1.09)

4. Secondary Outcome: Core Study: Mean Change From Baseline at Month 12 in Central Retinal Thickness of the Study Eye
Description: Retinal thickness was measured using Optical Coherence Tomography (OCT). The images were reviewed by a central reading center to ensure a standardized evaluation.
Time Frame: Baseline to Month 12
Population: The number analyzed is the Full Analysis Set, including patients with a value at both baseline and the Month 12 visit. Last Observation Carried Forward imputation was utilized.
Measure: Mean (Standard Deviation); unit: Micrometers
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser
Number analyzed (Participants) | 113 | 116 | 108
Micrometers
  Baseline | 427.1 (118.42) | 416.4 (119.91) | 412.4 (124.53)
  Value at Month 12 | 308.4 (112.26) | 288.2 (90.11) | 351.1 (139.91)
  Change from Baseline | -118.7 (115.07) | -128.3 (114.34) | -61.3 (132.29)

5. Secondary Outcome: Core Study: Mean Change From Baseline in Patient-reported Visual Functioning
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) was used to measure a patient's subjective assessment of vision-related quality of life. The 12 subscales in the VFQ-25 are general health, general vision, ocular pain, near activities, distance activities, social function, mental health, role difficulties, dependency, driving, color vision, and peripheral vision. The scores on the subscales were added together for a total score, which ranged from 0 to 100. A higher score indicated improvement in quality of life due to vision function.
Time Frame: Baseline to Month 12
Population: The number analyzed is the Full Analysis Set, including the number of patients with a value at both baseline and the Month 12 visit. Last Observation Carried Forward imputation was utilized.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser
Number analyzed (Participants) | 114 | 116 | 108
Units on a scale
  Baseline | 72.8 (16.91) | 74.1 (18.06) | 73.5 (18.18)
  Month 12 | 77.8 (19.19) | 79.5 (17.29) | 74.1 (18.80)
  Change from Baseline | 5.0 (12.97) | 5.4 (11.14) | 0.6 (12.56)

6. Primary Outcome: Extension Study: Percentage of Participants With Ocular Adverse Events (AEs) in the Study Eye in the 24 Month Extension Study
Description: Participants with ocular (occurring in the eye) serious adverse events (SAEs) and non-serious AEs in the study eye. The study eye is the eye that received the treatment. AEs are the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event is not considered to be related to study drug. A serious adverse event is defined as an event that is fatal or life-threatening, results in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, requires inpatient hospitalization or prolongation of existing hospitalization or is medically significant.
  Additional information about adverse events can be found in the Adverse Event section.
Time Frame: Extension baseline (Month 12 -end of core study) to Month 36 (end of extension study) [24 Months]
Population: Safety Population included all participants who entered the extension and who had at least one safety assessment in the extension study. Participants were grouped according to the treatment assigned in the Core study.
Measure: Number; unit: Percentage of participants
Groups:
- Laser With Ranibizumab in Extension; Laser Without Ranibizumab in Extension: Active laser photocoagulation treatment was administered on Day 1 and at intervals of at least 3 months, if deemed necessary by the evaluating physician. Patients also received monthly sham intravitreal injection in the study eye for 3 consecutive months. After the third injection, treatment was suspended if either one of the following criteria was met:
  Improvement in best corrected visual acuity (BCVA) could not be attributed to treatment at the last 2 visits, in the opinion of the investigator, or BCVA > 84 letters (approximate Snellen equivalent of 20/20) was observed at the last 2 last visits.
  Active/sham laser treatment was always administered before (sham) intravitreal injections. The minimum interval between the 2 treatments was 30 minutes.
  In the extension study at the investigator's discretion, patients received open-label ranibizumab 0.5 mg intravitreal injections once a month until stable vision was reached (a maximum of 24 injections) and could receive laser therapy.
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser With Ranibizumab in Extension | Laser Without Ranibizumab in Extension
Number analyzed (Participants) | 83 | 83 | 59 | 15
Percentage of participants
  Adverse Events | 56.6 | 56.6 | 52.5 | 40.0
  Serious Adverse Events | 2.4 | 1.2 | 1.7 | 0.0

7. Secondary Outcome: Extension Study: Percentage of Participants With Ocular Adverse Events (AEs) in the Study Eye in the 36 Months of the Core and Extension Studies
Description: as for outcome 6
Time Frame: Core baseline (Day 1 of the core study) to Month 36 (end of extension study) [36 months]
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser With Ranibizumab in Extension | Laser Without Ranibizumab in Extension
Number analyzed (Participants) | 83 | 83 | 59 | 15
Percentage of participants
  Adverse Events | 66.3 | 67.5 | 64.4 | 46.7
  Serious Adverse Events | 2.4 | 3.6 | 5.1 | 0.0

8. Secondary Outcome: Extension Study: Percentage of Participants With Non-Ocular Adverse Events (AEs) in the 36 Months of the Core and Extension Studies
Description: Participants with non-ocular (not occurring in the eye) serious adverse events (SAEs) and non-serious AEs. AEs are the appearance or worsening of of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event is not considered to be related to study drug. A serious adverse event is defined as an event that is fatal or life-threatening, results in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, requires inpatient hospitalization or prolongation of existing hospitalization or is medically significant.
  Additional information about Adverse Events can be found in the Adverse Event section.
Time Frame: Core baseline (Day 1 of the core study) to Month 36 (end of extension study) [36 Months]
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser With Ranibizumab in Extension | Laser Without Ranibizumab in Extension
Number analyzed (Participants) | 83 | 83 | 59 | 15
Percentage of participants
  Adverse Events | 83.1 | 81.9 | 84.7 | 73.3
  Serious Adverse Events | 36.1 | 37.3 | 42.4 | 13.3

9. Primary Outcome: Extension Study: Percentage of Participants With Non-Ocular Adverse Events (AEs) in the 24 Month Extension Study
Description: as for outcome 8
Time Frame: Extension baseline (Month 12 -end of core study) to Month 36 (end of extension study) [24 Months]
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser With Ranibizumab in Extension | Laser Without Ranibizumab in Extension
Number analyzed (Participants) | 83 | 83 | 59 | 15
Percentage of participants
  Adverse Events | 73.5 | 73.5 | 71.2 | 73.3
  Serious Adverse Events | 27.7 | 30.1 | 37.3 | 13.3

10. Secondary Outcome: Extension Study: Mean Change From Extension Study Baseline in Best Corrected Visual Acuity (BCVA) at Month 36
Description: Visual acuity (VA) was assessed on both eyes during every study visit using best correction determined from protocol refraction. VA measurements (number of letters correctly identified) were performed with the patient in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at a testing distance of 4 meters. An increase in the number of letters read correctly indicates improvement.
Time Frame: Extension baseline (Month12 -end of core study), Month 36 (end of extension study)
Population: Participants from the Safety Population that included all participants who entered the extension and who had at least one safety assessment in the extension study with data available for analyses. Participants were grouped according to the treatment assigned in the Core study.
Measure: Mean (Standard Deviation); unit: Letters
Groups:
- Active Laser: Active laser photocoagulation treatment was administered on Day 1 and at intervals of at least 3 months, if deemed necessary by the evaluating physician. Patients also received monthly sham intravitreal injection in the study eye for 3 consecutive months. After the third injection, treatment was suspended if either one of the following criteria was met:
  Improvement in best corrected visual acuity (BCVA) could not be attributed to treatment at the last 2 visits, in the opinion of the investigator, or BCVA > 84 letters (approximate Snellen equivalent of 20/20) was observed at the last 2 last visits.
  Active/sham laser treatment was always administered before (sham) intravitreal injections. The minimum interval between the 2 treatments was 30 minutes.
  In the extension study at the investigator's discretion, patients received open-label ranibizumab 0.5 mg intravitreal injections once a month until stable vision was reached (a maximum of 24 injections) and could receive laser therapy.
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Active Laser
Number analyzed (Participants) | 83 | 80 | 74
Letters | 0.1 (9.10) | -0.5 (9.19) | 3.7 (6.88)

11. Secondary Outcome: Extension Study: Mean Change From Core Study Baseline in Best Corrected Visual Acuity (BCVA) at Month 36
Description: as for outcome 10
Time Frame: Core baseline (Day 1 of the core study), Month 36 (end of extension study)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Active Laser
Number analyzed (Participants) | 83 | 83 | 74
Letters | 8.0 (10.09) | 6.7 (9.59) | 6.0 (9.35)

ADVERSE EVENTS:
Description: Safety Population included all randomized treated participants. Participants are grouped according to the treatment actually received in the Core Study.
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg + Laser | Laser With Ranibizumab in Extension | Laser Without Ranibizumab in Extension
Serious Adverse Events (participants affected / at risk) | 41/115 | 43/120 | 28/59 | 7/51
Other Adverse Events (participants affected / at risk) | 79/115 | 83/120 | 50/59 | 31/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=115) | Ranibizumab 0.5 mg + Laser (N=120) | Laser With Ranibizumab in Extension (N=59) | Laser Without Ranibizumab in Extension (N=51)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 3 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 4 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 3 | 1 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 4 | 3 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Spinocerebellar ataxia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Cataract (Fellow eye) (Eye disorders) | 2 | 1 | 1 | 0
Cataract (Study eye) (Eye disorders) | 0 | 3 | 2 | 0
Cataract subcapsular (Fellow eye) (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Corneal oedema (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Diabetic retinal oedema (Fellow eye) (Eye disorders) | 1 | 1 | 1 | 0
Lenticular opacities (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Vitreous adhesions (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Vitreous haemorrhage (Fellow eye) (Eye disorders) | 2 | 0 | 1 | 1
Vitreous haemorrhage (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Polyserositis (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Gas gangrene (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Mediastinitis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Eye injury (Fellow eye) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Eye injury (Study eye) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Eyelid injury (Study eye) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Periorbital haematoma (Study eye) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0
Body temperature decreased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Diabetic foot (Metabolism and nutrition disorders) | 2 | 0 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Urethral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 1 | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=115) | Ranibizumab 0.5 mg + Laser (N=120) | Laser With Ranibizumab in Extension (N=59) | Laser Without Ranibizumab in Extension (N=51)
Anaemia (Blood and lymphatic system disorders) | 2 | 6 | 3 | 1
Blepharitis (Fellow eye) (Eye disorders) | 1 | 1 | 3 | 1
Cataract (Fellow eye) (Eye disorders) | 10 | 12 | 7 | 5
Cataract (Study eye) (Eye disorders) | 9 | 17 | 9 | 4
Conjunctival haemorrhage (Study eye) (Eye disorders) | 9 | 13 | 0 | 0
Conjunctival hyperaemia (Study eye) (Eye disorders) | 9 | 8 | 5 | 2
Conjunctivitis (Fellow eye) (Eye disorders) | 4 | 6 | 3 | 1
Diabetic retinal oedema (Fellow eye) (Eye disorders) | 12 | 19 | 11 | 3
Diabetic retinal oedema (Study eye) (Eye disorders) | 7 | 6 | 3 | 1
Diabetic retinopathy (Fellow eye) (Eye disorders) | 4 | 6 | 4 | 2
Diabetic retinopathy (Study eye) (Eye disorders) | 3 | 8 | 3 | 2
Dry eye (Fellow eye) (Eye disorders) | 5 | 4 | 3 | 3
Dry eye (Study eye) (Eye disorders) | 5 | 4 | 3 | 3
Eye discharge (Study eye) (Eye disorders) | 4 | 6 | 1 | 1
Eye haemorrhage (Fellow eye) (Eye disorders) | 2 | 3 | 3 | 0
Eye haemorrhage (Study eye) (Eye disorders) | 2 | 3 | 3 | 0
Eye irritation (Study eye) (Eye disorders) | 3 | 2 | 3 | 0
Eye pain (Study eye) (Eye disorders) | 15 | 11 | 13 | 2
Eye pruritus (Study eye) (Eye disorders) | 3 | 3 | 5 | 1
Foreign body sensation in eyes (Study eye) (Eye disorders) | 5 | 8 | 2 | 0
Lacrimation increased (Study eye) (Eye disorders) | 3 | 6 | 5 | 0
Macular fibrosis (Study eye) (Eye disorders) | 2 | 2 | 5 | 0
Punctate keratitis (Fellow eye) (Eye disorders) | 1 | 6 | 0 | 0
Retinal aneurysm (Study eye) (Eye disorders) | 0 | 3 | 3 | 1
Retinal exudates (Fellow eye) (Eye disorders) | 7 | 3 | 3 | 1
Retinal exudates (Study eye) (Eye disorders) | 4 | 2 | 5 | 1
Retinal haemorrhage (Fellow eye) (Eye disorders) | 4 | 8 | 2 | 0
Vision blurred (Study eye) (Eye disorders) | 2 | 4 | 3 | 2
Visual acuity reduced (Fellow eye) (Eye disorders) | 4 | 3 | 3 | 2
Visual acuity reduced (Study eye) (Eye disorders) | 1 | 2 | 1 | 3
Vitreous haemorrhage (Study eye) (Eye disorders) | 1 | 1 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 6 | 5 | 2 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 3
Bronchitis (Infections and infestations) | 6 | 4 | 1 | 2
Influenza (Infections and infestations) | 12 | 8 | 8 | 5
Nasopharyngitis (Infections and infestations) | 18 | 21 | 15 | 8
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 4 | 5 | 4 | 1
Blood glucose increased (Investigations) | 1 | 3 | 3 | 1
Intraocular pressure increased (Fellow eye) (Investigations) | 3 | 6 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 8 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 3 | 1
Headache (Nervous system disorders) | 4 | 5 | 5 | 1
Renal failure (Renal and urinary disorders) | 1 | 2 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 4 | 1
Hypertension (Vascular disorders) | 15 | 11 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.